CLINICAL TRIAL: NCT06174324
Title: Visual Field Progression and RNFL Change After PreserFlo MicroShunt Implantation - a Prospective Cohort Study at the Ophthalmology Department Klinikum Klagenfurt
Brief Title: Visual Field Progression and RNFL Change After PreserFlo MicroShunt Implantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Klinikum Klagenfurt am Wörthersee (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Yosuf El-Shabrawi, Prim. Univ. Prof. Dr. Yosuf El-Shabrawi, Klinikum Klagenfurt am Wörthersee
Other Study IDs: S2021-29
Record Dates: First submitted 2023-09-26; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Glaucoma; Progression; Surgery
MeSH Terms: conditions — Glaucoma; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: PreserFlo Microshunt — The PreserFlo MicroShunt was invented to create a minimally invasive glaucoma drainage device, that comes close to the eye pressure reduction and safety profile of the current gold standard, the trabeculectomy. Reference: Pinchuk L, Riss I, Batlle JF, Kato YP, Martin JB, Arrieta E, Palmberg P, Parrish RK 2nd, Weber BA, Kwon Y, Parel JM. The development of a micro-shunt made from poly(styrene-block-isobutylene-block-styrene) to treat glaucoma. J Biomed Mater Res B Appl Biomater. 2017 Jan;105(1):211-221. doi: 10.1002/jbm.b.33525. Epub 2015 Sep 18. PMID: 26380916; PMCID: PMC5215625.

SUMMARY:
The trabeculectomy is the gold standard in glaucoma surgery, nevertheless often postoperative interventions have to be done. (1),(2) The PreserFlo MicroShunt (Santen, Osaka, Japan) implantation occurs without critical steps of trabeculectomy. (3) According to a study a 20% eye pressure reduction was achieved in 53.9% of patients one year after PreserFlo MicroShunt implantation and the risk of postoperative hypotony was clearly minimized. (4) It has been shown that after trabeculectomy there is a stable development of visual fields in the first 3 months after surgery and then, despite adequate intraocular pressure reduction, visual fields deteriorate. (5) At the Klinikum Klagenfurt structural and functional changes after PreserFlo MicroShunt Implantation shall be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with insufficient eye pressure control despite IOP (intraocular pressure)-lowering therapy
* Diagnosis of POAG (primary open angle glaucoma)
* Diagnosis of PEG (pseudoexfoliation glaucoma)
* Diagnosis of PDG (pigment dispersion glaucoma)
* Diagnosis of NTG (normal tension glaucoma)
* Agreement of patients to participate in the study

Exclusion Criteria:

* Previous glaucoma surgery
* Visual acuity of Nulla Lux
* Poor general condition
* Pregnancy
* Exudative macular degeneration

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with insufficient eye pressure control despite IOP-lowering therapy and the diagnosis of glaucoma
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2024-09-09 (Estimated); Study Completion 2024-09-09 (Estimated)

PRIMARY OUTCOMES:
Visual field progression (mean deviation, MD) 1 month postoperative, 3 months postoperative, 6 months and 12 months postoperative after PreserFlo MicroShunt Implantation. | Visual fields taken at baseline should be compared to visual fields 1 month postoperativ, 3 months postoperative and 1 year postoperative.
  Visual fields of patients at baseline preoperative and 1 month postoperative, 3 months postoperative, 6 months postoperative and 12 months postoperative should be compared.
RNFL (retinal nerve fiber layer) at baseline before sugery and changes after1 month, 3 months, 6 months and 12 months postoperative after PreserFlo MicroShunt Implantation will be evaluated. | The measurement of the nerve fiber index shall be done at baseline before surgery and 1 month, 3 months, 6 months and 12 months after surgery.
  The measurement of the nerve fiber will be compared at baseline before surgery to the values at 1 month, 3 months, 6 months and 12 months after surgery.
Intraocular pressure will be taken 1 month, 3 months, 6 months and 12 months after PreserFlo MicroShunt Implantation. | The intraocular pressure will be taken postoperative after one month, 3 months, 6 months and 12 months.
  The evaluation of the intraocular pressure shall be done 1 month, 3 months, 6 months and 12 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Yosuf El-Shabrawi, Principal Investigator — Klinikum Klagenfurt am Wörthersee
Locations (1):
- KlinikumKlagenfurt, Klagenfurt, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gedde SJ, Herndon LW, Brandt JD, Budenz DL, Feuer WJ, Schiffman JC; Tube Versus Trabeculectomy Study Group. Postoperative complications in the Tube Versus Trabeculectomy (TVT) study during five years of follow-up. Am J Ophthalmol. 2012 May;153(5):804-814.e1. doi: 10.1016/j.ajo.2011.10.024. Epub 2012 Jan 14. PMID 22244522
- [Background] Pinchuk L, Riss I, Batlle JF, Kato YP, Martin JB, Arrieta E, Palmberg P, Parrish RK 2nd, Weber BA, Kwon Y, Parel JM. The development of a micro-shunt made from poly(styrene-block-isobutylene-block-styrene) to treat glaucoma. J Biomed Mater Res B Appl Biomater. 2017 Jan;105(1):211-221. doi: 10.1002/jbm.b.33525. Epub 2015 Sep 18. PMID 26380916
- [Background] Baker ND, Barnebey HS, Moster MR, Stiles MC, Vold SD, Khatana AK, Flowers BE, Grover DS, Strouthidis NG, Panarelli JF; INN005 Study Group. Ab-Externo MicroShunt versus Trabeculectomy in Primary Open-Angle Glaucoma: One-Year Results from a 2-Year Randomized, Multicenter Study. Ophthalmology. 2021 Dec;128(12):1710-1721. doi: 10.1016/j.ophtha.2021.05.023. Epub 2021 May 27. PMID 34051211
- [Background] Chua J, Kadziauskiene A, Wong D, Asoklis R, Lesinskas E, Quang ND, Chong R, Tan B, Girard MJA, Mari JM, Crowston JG, Aung T, Schmetterer L. One year structural and functional glaucoma progression after trabeculectomy. Sci Rep. 2020 Feb 18;10(1):2808. doi: 10.1038/s41598-020-59792-9. PMID 32071369
- [Result] Rathi S, Andrews CA, Greenfield DS, Stein JD. Trends in Glaucoma Surgeries Performed by Glaucoma Subspecialists versus Nonsubspecialists on Medicare Beneficiaries from 2008 through 2016. Ophthalmology. 2021 Jan;128(1):30-38. doi: 10.1016/j.ophtha.2020.06.051. Epub 2020 Jun 26. PMID 32598949